CLINICAL TRIAL: NCT02094092
Title: L.Reuteri ProTectis DSM 17938 to Relieve Infant Colic and Its Effects on Infant Sleep Pattern & Maternal Mental Health. PRIC-SMM Trial
Brief Title: Role of ProTectis on Infant Colic and Its Effect on Infant Crying Time and Maternal Mental Health
Acronym: PRIC-SMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ferozsons Laboratories Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Parveen Akhtar, Head of Pediatric Department, Fauji Foundation Hospital, Ferozsons Laboratories Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FZSPBT001
Record Dates: First submitted 2014-03-13; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Infantile Colic; Infant Sleeping Habits; Maternal Mental Health.
Keywords: L.reuteri ProTectis DSM 17938; Infantile colic; Maternal mental health.; Infant crying/fussing; Edinburgh Postnatal Depression Scale (EPDS)
MeSH Terms: conditions — Colic | interventions — WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ProTectis drops (Placebo Comparator): Arm A.
  Interventions: Other: ProTectis drops (five drops per day) for 21 days
- Placebo drops (Placebo Comparator): Arm B
  Interventions: Other: Placebo drops (five drops per day) for 21 days

INTERVENTIONS:
Other: ProTectis drops (five drops per day) for 21 days
  Arms: ProTectis drops
Other: Placebo drops (five drops per day) for 21 days
  Arms: Placebo drops

SUMMARY:
This study will work on hypothetical assumption that compared to the arm supplemented with placebo (control) group; the L reuteri (intervention) group will lower daily crying/fussing time per 24 hours at one month post randomization. And that the L reuteri (intervention) group at 7, 14, 21, days and 1 week after the therapy cessation will have:

* Lower crying/fussing time per 24 hours.
* Relief from colic pain
* Longer sleep duration,
* Higher scores on a standardized measure of maternal mental health

DETAILED DESCRIPTION:
The present study is aimed to test the hypothesis that "modulating" the gut micro flora of colicky infants through the oral administration of Probiotic- ProTectis would not only decrease crying time related to infantile colic but will also improve sleeping habits of infant and consequently decrease/eradicate maternal mental stress.

1. This is a prospective, single center, Randomized, Double Blind, and Placebo Controlled Study. The study will be conducted according to GCP guidelines and in accordance with declaration of Helsinki. The protocol and informed consent will be approved by ethical committee of study center prior to initiation. Enrollment of infants in study will take place only after the procurement of written informed consent from parents.

Minimum 60 patients will be recruited and assessed over 1 week after treatment to characterize the pattern of product related adverse events (as per ICH- E1Guidelines criteria required for safety assessment for drugs intended for short term treatment). Personal and clinical data will be collected from CRF given to Investigator for a period of 3 weeks of treatment after the date of randomization and treatment initiation. Follow-up and causality assessment of medically significant events will also be undertaken.Study comprises of 5 total visits including Visit 1 that will be the recruitment, screening and treatment initiation visit. Clinical evaluation for patient eligibility will be assessed at this visit before final enrolment. Patient will be asked to come at day7 (visit 2), day14 (visit3), day21 (visit4), and a visit one week after visit 4(follow up visit 5) to monitor any change in treatment parameter and also to assess any AaDR. Any labs if required will be done at the discretion of investigator. Patient will be instructed to promptly report any unexplained side effects.

1. Study Analysis Upon completion of study duration, data will be analyzed to find out its effect on efficacy points set for concluding study results.

   For statistical analysis, Data will be entered and analyzed using SPSS version19. Some esoteric statistical test will be applied like percentages will be calculated for checking efficacy and for comparison we will apply paired t-test, also for graphical representation, we will make bar charts and pie charts.
2. Study Duration:

   Study is planned to be completed in 28 days after first enrollment. The visits after the screening/enrollment (V1) are scheduled at day 7(V2), 14(V3), 21(V4), 28(V5). Follow-Up visit 5:21day's treatment followed by one follow up visit one week after.

   2.The study physician will be examining infants at all visits. Parents will be encouraged to keep their infants in the study for follow-up visits even in cases of discontinuation of the study products.

   3. For our current study we measure the Parent's perception of colic severity by a 10-cm VAS in which a score of 0 indicated no pain and 10 indicated the worst pain. For assessment of Parental/family quality of life, 0 indicated no effect and 10 indicated a very good effect. Parents will be instructed how to use the VAS scale prior to the study. At Screening V1, V4 and Follow Up V5 Visits 0 -------1--------2--------3--------4--------5--------6---------7--------8--------9------ 10 Poor fair good very good excellent

   3. Edinburgh Postnatal Depression Scale (EPDS): Postnatal Depression Scale (EPDS) is a valuable and efficient way of identifying patients at risk for "perinatal" depression. The EPDS is easy to administer and has proven to be an effective screening tool. Mothers who score above 13 are likely to be suffering from a depressive illness of varying severity. The EPDS score should not override clinical judgment. A careful clinical assessment should be carried out to confirm the diagnosis. The scale indicates how the mother has felt during the previous week. In doubtful cases it may be useful to repeat the tool after 2 weeks. The scale will not detect mothers with anxiety neuroses, phobias or personality disorders. The mother is asked to check the response that comes closest to how she has been feeling in the previous 7 days not just how she feels today.

   4. It is planned to enrolled at-least 60 patients in this study.

   5. All patients have the right to withdraw at any point during treatment without prejudice. The investigator can discontinue any patient at any time if medically necessary. It will be documented whether or not each patient completed the clinical study. If for any patient study treatment or observations were discontinued, the reason will be recorded and the sponsor should be notified promptly. Reasons that a patient may discontinue participation in a clinical study are considered to constitute one of the following:
   * Adverse event(s), including an event resulting in death
   * Abnormal labs result(s)
   * Unsatisfactory therapeutic effect
   * Protocol violation
   * Patient withdrew consent
   * lost to follow-up
   * Administrative problems

     6. It is imperative to obtain complete follow-up data for all patients whether or not they receive their assigned treatment or have discontinued study drug. Every attempt should be made to collect follow-up information except for those patients who specifically withdraw consent release of such information.

     7. Oil based L reuteri ProTectis DSM 17938 (five drops per day=108CFU) for 21 days will be used as study product in intervention group. The placebo (to be provided by BioGaia AB Stockholm Sweden) will be an oil based malt dextrose formulation having the same Appearance, Packaging and taste as that of intervention. Both placebo and study product will be labeled with
   * Randomization number
   * Batch number
   * Expiry date
   * And the statement "For clinical trial use only".

   Arm A: ProTectis drops (five drops per day) for 21 days. Arm B: Placebo drops (five drops per day) for 21 days. Sponsor will provide the study medication for the whole study period.

   8. As per the available clinical data on Lactobacillus reuteri DSM 17938 till date, no drug / food interaction of clinical significance has been reported. However it is important to keep the sensitivity profile of this Probiotic bacterium to antibiotics.

   9. The treatment, dosage and period of administration for study drug administered must be documented. A monitor will review patient source documents and drug accountability records to assess treatment compliance on an on-going basis during site visits.

   10. Investigational product should be stored in a secure area. It is the responsibility of the investigator to ensure that investigational product is only dispensed to study patients. The investigational product must be dispensed only from official study site by authorized personnel. It is the responsibility of the investigator to ensure that a current record of investigational product disposition is maintained at study site. Upon completion or termination of the study, all unused and/or partially used investigational product must be returned to the sponsor.

   11. This study will be conducted in compliance with the (ICH) GCP guidelines and with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* All infants (Full term with gestational age > 37 weeks and < 41 weeks) aged <3 months with infantile colic (defined as crying episodes lasting 3 or more hours/day and occurring at least 3 days/week within 7 days prior to enrollment)
* Infants who were exclusively or predominantly (>50%) breastfed/fed on Fresh Milk i.e.; cow milk/buffalo/tetra pack.

Exclusion Criteria:

* Acute or chronic illness
* Gastrointestinal disorders
* Use of any antibiotics and/or probiotic pharmaceutical products within 7 days prior to the study.
* Infants taking Probiotic containing infant formula milks.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The treatment success (defined as the percentage of children achieving a reduction in the daily average crying time 50% during the study) | Day 28
Change in the duration of crying (minutes per day). | Base line, day 7, day 14, day 21 & day 28

SECONDARY OUTCOMES:
A reduction in the daily average crying time, to <3 h/d. | Day 21
Change in Infant sleep duration in (minutes/day) | Baseline, day 7, day 14, day 21& day 28
Change in Maternal mental health scores. | Baseline, day 21 & day 28

OTHER OUTCOMES:
Persistence of infantile colic after the intervention. | Day 28
Change in the Parental perceptions of colic severity | Baseline, day 7, day 14, day 21 & day 28
Change in the Parental/ family quality of life | Baseline, day 21 & day 28

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Akhter, Dr., Principal Investigator — Fauji Foundation Hospital
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan